CLINICAL TRIAL: NCT01912170
Title: Effect of Omega-3 Fatty Acids on Insulin Sensitivity in Chinese Gestational Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DUOLI_GD
Record Dates: First submitted 2013-07-27; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Gestational Diabetes
Keywords: omega-3 fatty acid; gestational diabetes; insulin sensitivity
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Fish Oils; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- fish oil (Experimental): Patients will receive fish oil capsules, at a dose of 2g/day. Each 1g capsule will contain 220mg of EPA and 170mg of DHA
  Interventions: Dietary Supplement: Fish oil
- Flaxseed Oil (Experimental): Patients will receive flaxseed oil capsule, at a dose of 2g/day. Each 1g capsule will contain 550mg of ALA
  Interventions: Dietary Supplement: Flaxseed oil
- Placebo Supplementation (Placebo Comparator): Patients will receive corn oil in the capsules at the same dose as fish oil. The corn oil will appear identical in size and color to the fish oil

INTERVENTIONS:
Dietary Supplement: Fish oil
  Arms: fish oil
Dietary Supplement: Flaxseed oil
  Arms: Flaxseed Oil

SUMMARY:
This study is to examine the change of fasting insulin, glucose, insulin sensitivity and related traits in response to the 14 wk treatment of omega-3 fatty acids, including fish oil (n=25) and flaxseed oil(n=25), in Chinese gestational diabetic patients. Corn oil(n=25), rich in omega-6 fatty acids, will be selected as a controlled oil. The intervention will start from the third trimester of these pregnant women and finish at the 4wk after the birth of their children. The investigators hypothesize that omega-3 fatty acids could improve insulin sensitivity and glucose metabolism in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 1)gestational diabetes 2) female, <40 years old 3)willing to participant in the trial

Exclusion Criteria:

* 1）type 1 diabetes or type 2 diabetes before pregnancy 2）Deny to sign the informed consent 3）Family history of hypertriglyceridemia or fasting triglyceride>4.56 mmol/L 4）Have severe liver disease, kidney disease or cancer 5)Participating in the other clinical trial within 30 days 6)Other diseases or conditions, for which the doctor of the patients do not agree his or her participating

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
fasting glucose | 14 weeks
Fasting insulin | 14 weeks

SECONDARY OUTCOMES:
birth weight, length of children | 10 weeks

OTHER OUTCOMES:
blood lipids, inflammatory markers | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jiaxing Women's and Children's Hospital, Jiaxing, Zhejiang, China